CLINICAL TRIAL: NCT05299918
Title: Diabetic Neuropathy Rapid Screening Test in Turkish Patients With Type 2 Diabetes Sudoscan
Brief Title: Diabetic Neuropathy Rapid Screening Test in Turkish Patients With Type 2 Diabetes: Sudoscan
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Calikoglu, MD, PhD; Academician; Principle Investigator, Istanbul University
Other Study IDs: 2014/495
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Neuropathy Autonomic; Cardiac Autonomic Neuropathy; Type2Diabetes; Diabetic Neuropathy Peripheral; Diabetic Neuropathies
Keywords: SUDOSCAN; Cardiac Autonomic Neuropathy; Neuropathy Autonomic; Diabetic Neuropathy Peripheral; Type2Diabetes
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuropathy is a frequently observed complication occurring in 60-70% of diabetic patients throughout their lives. In addition, neuropathy is a severe disease that progresses insidiously; its diagnosis can be delayed due to the absence of clinical findings, affects the quality of life, and increases mortality and morbidity. Up to 50% of patients with diabetic peripheral neuropathy (DPN) may be asymptomatic. Typically, DPN progresses in the form of chronic, symmetrical, and progressive sensorimotor polyneuropathy. The five-year mortality rate of individuals with diabetes with autonomic neuropathy is three times higher than those without. The diagnosis of clinical neuropathy is usually made by the symptoms, the vibration sensation with the diapason, and the tactile sensation tests. Although diapason and monofilament tests are easy, they are qualitative tests that the patient must be careful and coordinate with. Biothesiometry or Semmes-Weinstein monofilament tests cannot examine autonomous involvement. Cardiovascular autonomic neuropathy tests based on heart rate variability (HRV), on the other hand, can be affected by factors such as age, body position, cigarette-coffee consumption, blood pressure, exercise, heart rate, and respiratory rate. An easy and fast diagnostic method may be more helpful in diagnosing peripheral and autonomic neuropathy.

Distal small-fiber polyneuropathy can be detected by measuring sweat function using Sudoscan, a rapid, non-invasive, and quantitative method. This measurement method is based on the electrochemical reaction between sweat chlorides and stainless steel electrodes that come into contact with the palms of the hands and soles of the feet. Results are provided as a Diabetic Autonomic Neuropathy (DAN) score based on conductances (micro siemens, μS) and conductivity values for the hands and feet (right and left sides). SUDOSCAN can detect distal small-fiber polyneuropathy with >75% sensitivity. SUDOSCAN can be considered a robust method for detecting sudomotor dysfunction and is used for clinical and research purposes.

In the American Diabetes Association (ADA) consensus statement, sudomotor functions are mentioned in the early diagnosis of autonomic neuropathy in people with diabetes.

This study aimed to evaluate the effectiveness of this method in clinical applications by comparing sudomotor test results with other conventional measurement methods in the evaluation of diabetic peripheral and cardiac neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* The ability to give informed consent
* Male or female persons >18 years of age with a diagnosis of type 2 DM (WHO criteria)

Exclusion Criteria:

* <18 years of age
* Participants with type 1 diabetes
* Ongoing cancer treatment or other concurrent illness that will make the patient unable to attend the study at the discretion of the investigator
* Pregnant or breastfeeding participants
* Participants with atrial fibrillation, atrial flutter, or pacemakers will not be subjected to cardiac autonomic neuropathy measurements.
* Participants with toe or foot amputations or foot ulcer
* vitamin B12 deficiency and other causes of peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was selected among adult type 2 diabetes patients under control at Istanbul University Istanbul Medical Faculty Diabetes Polyclinic between July 2014 and July 2015. The 437 patients included studying were the ages of 18 and older.
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Peripheral Neuropathy assesed by sudoscan | 15.07.2014 to15.07.2015
  Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance (µS) in feet
Peripheral Neuropathy assesed by sudoscan | 15.07.2014 to15.07.2015
  Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance (µS) in hands
Peripheral Neuropathy assesed by Monofilament | 15.07.2014 to15.07.2015
  Neuropathy assesed by Monofilament Light touch with 10 g monofilament
Peripheral Neuropathy assesed by Douleur Neuropathique 4 Questions (DN4) | 15.07.2014 to15.07.2015
Peripheral Neuropathy assesed by diapason | 15.07.2014 to15.07.2015
  Neuropathy assessed by diapason Light touch with 128 Hz diapason
Cardiac Autonomic Neuropathy assesed by electrocardiogram (ECG) | 15.07.2014 to15.07.2015
  The expiration/inspiration (E/I) ratio was calculated by dividing the mean of the longest RR interval during expiration by the mean of the shortest RR interval during inspiration while the patient was lying quietly and breathing deeply with an electrocardiogram recording the heart rate change. This ratio is considered ≥ 1.21 normal, between 1.11-1.20 borderline, and ≤ 1.1 abnormal.
Peripheral Neuropathy assesed by NC-Stat (Neurometrix) | 15.07.2014 to15.07.2015
  In the evaluation of Neurometric Measurement; normal limits are >4 microvolts and >40 second meters
Cardiac Autonomic Neuropathy assesed by Othostatic BP change | 15.07.2014 to15.07.2015
  The blood pressure is measured using a standard sphygmomanometer while the subject is lying down again after standing up. The difference in systolic blood pressure is taken to measure postural blood pressure change. The measured blood pressure difference is considered normal if ≤10 mmHg, borderline between 11-29 mmHg, and abnormal if ≥30 mmHg.

REFERENCES:
- [Result] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Result] Gin H, Baudoin R, Raffaitin CH, Rigalleau V, Gonzalez C. Non-invasive and quantitative assessment of sudomotor function for peripheral diabetic neuropathy evaluation. Diabetes Metab. 2011 Dec;37(6):527-32. doi: 10.1016/j.diabet.2011.05.003. Epub 2011 Jun 28. PMID 21715211
- [Result] Mayaudon H, Miloche PO, Bauduceau B. A new simple method for assessing sudomotor function: relevance in type 2 diabetes. Diabetes Metab. 2010 Dec;36(6 Pt 1):450-4. doi: 10.1016/j.diabet.2010.05.004. Epub 2010 Aug 23. PMID 20739207
- [Result] Ewing DJ, Martyn CN, Young RJ, Clarke BF. The value of cardiovascular autonomic function tests: 10 years experience in diabetes. Diabetes Care. 1985 Sep-Oct;8(5):491-8. doi: 10.2337/diacare.8.5.491. PMID 4053936
- [Result] Casellini CM, Parson HK, Richardson MS, Nevoret ML, Vinik AI. Sudoscan, a noninvasive tool for detecting diabetic small fiber neuropathy and autonomic dysfunction. Diabetes Technol Ther. 2013 Nov;15(11):948-53. doi: 10.1089/dia.2013.0129. Epub 2013 Jul 27. PMID 23889506
- [Result] Yajnik CS, Kantikar VV, Pande AJ, Deslypere JP. Quick and simple evaluation of sudomotor function for screening of diabetic neuropathy. ISRN Endocrinol. 2012;2012:103714. doi: 10.5402/2012/103714. Epub 2012 Jul 9. PMID 22830040
- [Result] Grandinetti A, Chow DC, Sletten DM, Oyama JK, Theriault AG, Schatz IJ, Low PA. Impaired glucose tolerance is associated with postganglionic sudomotor impairment. Clin Auton Res. 2007 Aug;17(4):231-3. doi: 10.1007/s10286-007-0426-z. Epub 2007 Aug 23. PMID 17717720
- [Result] Low VA, Sandroni P, Fealey RD, Low PA. Detection of small-fiber neuropathy by sudomotor testing. Muscle Nerve. 2006 Jul;34(1):57-61. doi: 10.1002/mus.20551. PMID 16718689
- [Result] Unal-Cevik I, Sarioglu-Ay S, Evcik D. A comparison of the DN4 and LANSS questionnaires in the assessment of neuropathic pain: validity and reliability of the Turkish version of DN4. J Pain. 2010 Nov;11(11):1129-35. doi: 10.1016/j.jpain.2010.02.003. Epub 2010 Apr 24. PMID 20418179
- [Result] Selvarajah D, Cash T, Davies J, Sankar A, Rao G, Grieg M, Pallai S, Gandhi R, Wilkinson ID, Tesfaye S. SUDOSCAN: A Simple, Rapid, and Objective Method with Potential for Screening for Diabetic Peripheral Neuropathy. PLoS One. 2015 Oct 12;10(10):e0138224. doi: 10.1371/journal.pone.0138224. eCollection 2015. PMID 26457582